CLINICAL TRIAL: NCT06935318
Title: Effects of an 11-Week High Functional Resistance Training Program on Indices of Arterial Stiffness
Brief Title: Effects of High Functional Resistance Training Program on Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salisbury University (Other)
Responsible Party: Principal Investigator, Timothy Werner, Professor, Salisbury University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: #1
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Training Study
Keywords: pulse wave velocity; beta-stiffness index; central arterial blood pressure; CrossFit training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental)
  Interventions: Other: Exercise
- Control Group (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — The exercise group performed an 11-week high-functional resistance program in a group training format. They trained 3-4 days a week following nationally assigned workouts
  Arms: Exercise Group
Other: Control — Did not participate in exercise related activities for the duration of the study period.
  Arms: Control Group

SUMMARY:
Study examined the effects of CrossFit training on blood vessels. The results indicate long term CrossFit training does not harm blood vessel function.

DETAILED DESCRIPTION:
Arterial stiffness is a systemic loss of elastic properties that significantly augment cardiovascular disease risk in adults. Chronic aerobic and anaerobic exercise activity has consistently been shown to attenuate or not affect markers of arterial stiffness in adults with chronic disease and otherwise healthy adults. Chronic high functional resistance training's effect on vascular compliance is less understood. The study aimed to determine the impact of a chronic high functional resistance training program on pulse wave velocity and beta-stiffness index. Accordingly, participants (18-40 years old) were placed in a non-randomized fashion into high functional resistance training (HIB) group (n = 9; >6 months of CrossFit experience; 4 female) or control (CON) group (n = 8; < 6 months of exercise experience; 6 female). Participants in the HIB group trained at the same local facility 4 -5 days a week, utilizing the same training program. CON group refrained from exercise during the study period. Body composition, 1,000-meter rowing test, deadlift 1 repetition maximum (1 RM), hemodynamic assessments, and vascular compliance were assessed at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* body weight stability with no more than ± 2.5 kg fluctuations in last six month

Exclusion Criteria:

* hypertension
* heart disease
* cancer
* diabetes
* renal disease
* hepatic disorders
* history of tobacco use.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-29 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity | From enrollment to the end of treatment at 11 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Salisbury University, Salisbury, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Garcia-Mateo P, Garcia-de-Alcaraz A, Rodriguez-Perez MA, Alcaraz-Ibanez M. Effects of Resistance Training on Arterial Stiffness in Healthy People: A Systematic Review. J Sports Sci Med. 2020 Aug 13;19(3):444-451. eCollection 2020 Sep. PMID 32874096